CLINICAL TRIAL: NCT07202858
Title: Validation of the STARZ Score for Early Prediction of Neonatal Acute Kidney Injury in Assuit University Children Hospital
Brief Title: Validation of STARZ Score for Early Neonatal AKI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menna Allah Talaat Mahmoud, Validation of the STARZ score in early prediction of neonatal acute kidney injury in Assuit university children hospital, Assiut University
Other Study IDs: STARZ-AKI-NEO-Assiut
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury; Kidney Diseases; Newborn
Keywords: Neonatal Acute Kidney Injury; STARZ Score; NICU
MeSH Terms: conditions — Acute Kidney Injury; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neonatal acute kidney injury (AKI) is a common complication in the NICU, associated with high morbidity and mortality. Prematurity, low birthweight, sepsis, asphyxia, congenital heart disease, and nephrotoxic drugs are major risk factors. Early diagnosis is challenging as serum creatinine lacks sensitivity. The STARZ score, a composite clinical-laboratory tool, has shown high accuracy for predicting early neonatal AKI. This study aims to validate the STARZ score in neonates admitted to Assiut University Children's Hospital for early identification of AKI and improved clinical outcomes."

DETAILED DESCRIPTION:
Neonatal acute kidney injury (AKI) is a frequent and serious complication in the neonatal intensive care unit (NICU), with incidence rates ranging from 6% to 24% and reaching up to 70% in high-risk populations depending on diagnostic criteria. Prematurity, low birthweight, sepsis, perinatal asphyxia, congenital heart disease, respiratory distress, shock, and exposure to nephrotoxic medications are established risk factors. Neonatal AKI is associated with increased mortality, prolonged hospitalization, and long-term renal complications, including chronic kidney disease.

Traditional diagnostic tools, such as serum creatinine, are limited by delayed changes and poor sensitivity in neonates. Risk stratification models offer an opportunity for earlier detection and proactive intervention. The STARZ score is a composite risk assessment tool incorporating clinical and laboratory parameters, and has demonstrated high predictive accuracy in previous studies, with sensitivity above 85% and specificity around 90% for early neonatal AKI.

This prospective study at Assiut University Children's Hospital aims to validate the STARZ score for predicting neonatal AKI within the first 7 days of NICU admission. The study will assess its predictive performance compared with conventional criteria, evaluate its role in risk stratification and guiding timely interventions, and examine the potential benefits in terms of cost-effectiveness and healthcare resource utilization.

ELIGIBILITY:
* Neonates admitted to the NICU within 48 hours of birth.
* Gestational age ≥ 28weeks.
* Birth weight ≥ 1000grams.
* Neonates with clinical indications necessitating laboratory investigations relevant to kidney function monitoring as part of standard care.
* Parental or guardian consent obtained for study participation.

Exclusion Criteria:

* Neonates with known congenital renal anomalies diagnosed antenatally or postnatally.

  * Neonates with chromosomal abnormalities or genetic syndromes affecting renal function.
  * Neonates discharged, transferred, or deceased within 24 hours of admission.
  * Neonates with incomplete medical records or missing key laboratory data

Ages: 0 Hours to 28 Days | Sex: All
Age Groups: Child
Study Population: Neonates admitted to the neonatal intensive care unit (NICU) at Assiut University Children's Hospital within the first 24 hours of life. Both preterm and term neonates will be included. Participants will be evaluated for the risk of developing acute kidney injury (AKI) using the STARZ score during the first 7 days of admission.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Predictive accuracy of STARZ score for early neonatal AKI | Within the first 7 days of NICU admission
  Validation of the STARZ risk stratification score for identifying neonates at risk of AKI within the first 7 days of NICU admission

SECONDARY OUTCOMES:
Comparison of STARZ score with conventional AKI markers | Within the first 7 days of NICU admission
  Evaluate sensitivity, specificity, and predictive values of STARZ score versus serum creatinine and urine output

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhooria GS, Nautiyal A, Wazir S, Agrawal G, Tiwana A, Bajaj N, Gupta NP, Mirgunde S, Sahoo J, Balachandran B, Afzal K, Shrivastava A, Bagla J, Krishnegowda S, Konapur A, Soni K, McCulloch M, Bunchman T, Sethi SK, Raina R. Validation of the STARZ neonatal acute kidney injury risk stratification score in an independent prospective cohort. J Neonatal Perinatal Med. 2022;15(4):777-785. doi: 10.3233/NPM-221044. PMID 36189502
- [Background] Gupta S, Gaur BK, Jain R, Singh RR. Incidence, Risk Factors, and Outcomes of Acute Kidney Injury in Preterm Neonates Hospitalized in the Neonatology Unit, North India: A Single-center Experience. Saudi J Kidney Dis Transpl. 2023 Nov 1;34(6):592-601. doi: 10.4103/sjkdt.sjkdt_264_23. Epub 2024 May 9. PMID 38725209